CLINICAL TRIAL: NCT01683110
Title: An Open-Label, Expanded Access Study of Cabozantinib (XL184) in Subjects With Unresectable, Locally Advanced, or Metastatic Medullary Thyroid Cancer
Brief Title: Expanded Access of Cabozantinib in Medullary Thyroid Cancer
Status: Approved for marketing | Type: Expanded Access
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Other Study IDs: XL184-209
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Medullary Thyroid Cancer
MeSH Terms: conditions — Carcinoma, Medullary | interventions — cabozantinib

INTERVENTIONS:
Drug: cabozantinib

SUMMARY:
The objective of this study is to provide access to cabozantinib for eligible subjects with medullary thyroid cancer (MTC) pending approval of Exelixis' New Drug Application (NDA) by the FDA and commercial availability of cabozantinib.

ELIGIBILITY:
Inclusion Criteria:

* The subject has histologically confirmed diagnosis of MTC that is unresectable, locally advanced, or metastatic
* The subject has documented progressive disease (PD) as determined by the investigator
* The subject has been previously treated with available standard therapy for unresectable, locally advanced, or metastatic MTC; or other currently available therapy is considered inappropriate for the subject as determined by the investigator
* The subject has Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* The subject has adequate organ and marrow function
* The subject is capable of understanding and complying with the protocol requirements and has signed the informed consent document
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 3 months after the last dose of cabozantinib received as part of this study, even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control.

Exclusion Criteria:

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (eg, antibodies) within 4 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of cabozantinib
* The subject has previously been enrolled in a clinical trial evaluating cabozantinib including placebo-controlled trials in which the subject may not have been treated with cabozantinib
* The subject has received radiation therapy:

  1. to the thoracic cavity, abdomen, or pelvis within 12 weeks before the first dose of study treatment , or has ongoing complications or is without complete recovery and healing from prior radiation therapy
  2. to bone or brain metastasis within 14 days before the first dose of cabozantinib
  3. to any other site(s) within 28 days before the first dose of cabozantinib
* The subject has received radionuclide treatment within 6 weeks before the first dose of cabozantinib
* The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lifes of the compound or active metabolites, whichever is longer, before the first dose of cabozantinib
* The subject has received any other type of investigational agent within 28 days before the first dose of cabozantinib
* The subject has not recovered to baseline or CTCAE ≤ Grade 1 from toxicity due to all prior therapies except alopecia and other clinically non-significant side effects
* The subject has active brain metastases or epidural disease (certain exceptions apply)
* The subject requires chronic concomitant treatment of strong CYP3A4 inducers (eg, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St. John's Wort)
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (eg, clopidogrel). Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic low molecular weight heparin are permitted
* The subject has experienced any of the following:

  1. clinically-significant GI bleeding within 6 months before the first dose of cabozantinib
  2. hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood within 3 months before the first dose of cabozantinib
  3. any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of cabozantinib
* The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has radiographic evidence of tumor in contact with, invading or encasing any major blood vessel
* The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness (which may include certain cardiac disorders, certain gastrointestinal disorders, and major surgeries)
* The subject is unable to swallow capsules
* The subject is pregnant or breastfeeding
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* The subject has had another diagnosis of malignancy, requiring systemic treatment, within two years before the first dose of cabozantinib, unless that malignancy has been treated with curative intent and the subject is taking no other anti-cancer therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford, California
  - Boston, Massachusetts
  - Detroit, Michigan
  - Portland, Oregon
  - Philadelphia, Pennsylvania